CLINICAL TRIAL: NCT03213899
Title: Association Between Malnutrition and Hospital Mortality and Duration of Intensive Care Unit Admission in the Critically Ill: a Prospective Singapore Cohort Study
Brief Title: Association Between Malnutrition and Clinical Outcomes in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: JurongHealth (Other Government)
Collaborators: Flinders University (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/00878/2
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Critical Illness; Malnutrition
Keywords: Subjective Global Assessment; Nutritional Status; Hospital Mortality; Length of Stay; Malnutrition
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have demonstrated the direct associations between malnutrition and hospital mortality as well as the length of stay in critically ill patients. However, the validity of these results may be limited by inappropriate diagnoses of malnutrition, small sample size, possible treatment bias, and sub-optimal statistical adjustment. This study aimed to further examine the aforementioned associations by addressing these limitations.

DETAILED DESCRIPTION:
Design:

* Prospective cohort study

Setting:

* 35-bedded integrated intensive care/ high dependency unit in Ng Teng Fong General Hospital. Patients' status can be changed between ICU-status and HD-status within the same ICU-/ HD-bed

Participants:

* All adult patients who will be admitted to the unit between August-2015 to October-2016 for ≥ 24 hours

Intervention:

Nil. Given the observational nature of this study, no attempt will be made to standardize care, including nutritional practices.

Measurement:

* As per routine care, a validated nutritional assessment tool [7-point Subjective Global Assessment (7-point SGA)] will be used to determine patients' nutritional status within 48 hours of ICU admission
* The primary outcomes will be hospital mortality and ICU length of stay. To measure hospital mortality, all patients will be followed until hospital discharge or death for up to one year after ICU admission. For ICU length of stay (in days), duration will be measured from the date of the first ICU admission to the date of the first change in ICU-status to HD-status or discharge to the general ward

Analysis:

* Modified Cox regression model with robust variance and logistic regression will be used to determine the associations between nutritional status and hospital mortality. Analyses will be conducted in two ways: 1) presence versus absence of malnutrition, and 2) dose-dependent association for each 1-point decrease in the 7-point SGA
* Multiple linear regression will be applied to determine the associations between nutritional status and ICU length of stay

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old who had ≥ 24 hours length of stay in the ICU
* received a nutrition assessment (7-point SGA) from a dietitian within 48 hours of admission to the ICU

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients ≥ 18 years old who had ≥ 24 hours length of stay in the ICU, and received a nutrition assessment (7-point SGA) from a dietitian within 48 hours of admission to the ICU.
Sampling Method: Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | Up to one year after admission to the ICU
  Death during hospitalization
ICU length of stay | From the date of the first ICU admission to the date of the first change in ICU-status to HD-status or discharge to the general ward, for up to one year after admission to the ICU
  Duration of the first intensive care unit admission

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lew CCH, Yandell R, Fraser RJL, Chua AP, Chong MFF, Miller M. Association Between Malnutrition and Clinical Outcomes in the Intensive Care Unit: A Systematic Review [Formula: see text]. JPEN J Parenter Enteral Nutr. 2017 Jul;41(5):744-758. doi: 10.1177/0148607115625638. Epub 2016 Feb 2. PMID 26838530